CLINICAL TRIAL: NCT03434418
Title: A Single Arm Phase II Study Osimertinib in Patients With Stage 4 Non-small Cell Lung Cancer With Uncommon EGFR Mutations
Brief Title: A Study Osimertinib in Patients With Stage 4 Non-small Cell Lung Cancer With Uncommon EGFR Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00088376
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: EGFR Mutation; osimertinib; exon 18 G719X; exon 20 S7681; exon 21 L861Q
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- osimertinib (Experimental)
  Interventions: Drug: osimertinib

INTERVENTIONS:
Drug: osimertinib — 80 mg oral administration daily
  Other Names: Tagrisso

SUMMARY:
This is a research study to find out if a drug called, osimertinib, is safe and effective in treating advanced Non-Small Cell Lung Cancer (NSCLC) by targeting the treatment of epidermal growth factor receptor (EGFR) mutation exon 18 G719X, exon 20 S7681, or exon 21 L861Q. Patients on the study will not have had previous tyrosine kinase inhibitor (TKI) treatment.

DETAILED DESCRIPTION:
This is a research study to find out if a drug called, osimertinib, is safe and effective in treating advanced Non-Small Cell Lung Cancer (NSCLC) by targeting the treatment of epidermal growth factor receptor (EGFR) mutation exon 18 G719X, exon 20 S7681, or exon 21 L861Q. Patients on the study will not have had previous tyrosine kinase inhibitor (TKI) treatment.

Patients who have one of the following EGRF mutations: exon 18 G719X, exon 20 S7681, or exon 21 L861Q) may be eligible to participate in this study. If enrolled into the study, the study team will give the patient a supply of the study drug, osimbertinib (80 mg) to take at home. The patient will be asked to take the study drug by mouth on days 1-28 of each study cycle. As part of this study, the patient will have blood samples other tests, exams and procedures done for study purposes and their standard of care. Patient participation in the study will last for up to 2 years after completion of the last dose of the study drug or until your condition worsens or intolerable adverse events as deemed by the study doctor.

There are possible patient risks to this study that include but are not limited to diarrhea, changes to the lining of the mouth (e.g. ulcers), rash, dry skin, itching, and nail infections.

ELIGIBILITY:
Inclusion Criteria:

* EGFR mutations as performed on a CLIA certified laboratory demonstrating EGFR exon 18 G719X, exon 20 S768I, or exon 21 L861Q. Patients with compound (also referred to as multiple mutations) will be eligible provided the NSCLC demonstrates one of these mutations).
* Histological or cytological confirmation diagnosis of Stage 4 NSCLC.
* Measurable disease by RECIST 1.1 (please refer to appendix 4)
* The following laboratory values obtained ≤ 14 days prior to study initiation.
* Hematology: ANC ≥ 1, 500 / ml, platelet count, ≥ 100,000 / ml, hemoglobin ≥ 9.0 g / dl
* Hepatic:ALT or ALT < 2.5 times ULN if no demonstrable liver metastases or <5 times ULN in the presence of liver metastases
* Total bilirubin < 1.5 times ULN if no liver metastases or < 3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases
* Renal: Cockcroft-Gault calculated creatinine clearance of ≥ 45 ml/min or creatinine ≤1.5 x ULN
* Have normal QT interval on ECG evaluation QT corrected of ≤ 450 ms in males or ≤ 470 ms in females obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine-derived QTc value
* Cardiac ejection fraction of ≥ 45%
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or1
* Negative pregnancy test done ≤7 days (or per institutional policy) prior to treatment, for women of childbearing potential only. Female must use highly effective contraceptive measures, and must have a negative pregnancy test or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:
* Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
* Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
* Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* Male subjects must be willing to use barrier contraception
* Age ≥ 18 years
* Provision of written informed consent prior to any study-specific procedures

Exclusion Criteria:

* Prior therapy with EGFR TKI therapy
* Greater than 2 lines of prior systemic therapy for metastatic non-small cell lung cancer.
* Any cytotoxic chemotherapy or other anticancer drugs from previous treatment regimen or clinical study within 14 days of first dose of study drug.
* Treatment with an investigational drug within 5 half-lives of the compound
* Other active malignancy ≤ 2 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix. NOTE: If there is a history of prior malignancy, patients must not be receiving other specific treatment (i.e. hormonal therapy) for their cancer
* Prior radiotherapy ≤ 14 days
* Untreated symptomatic brain metastases (treated brain metastases are allowed provided > 14 days have elapsed from completion of radiotherapy and patient is neurologically stable as assessed by treating physician).
* Malabsorption syndrome, refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib
* Detection of concurrent EGFR mutation with exon 20 T790M, exon 19 deletion, exon 21 L858R mutation or exon 20 insertion. Patients with compound (also referred to as multiple mutations) will be excluded if the molecular testing includes one of these mutations.
* Active pregnancy or breast-feeding: Pregnant women are excluded from this study because the effects of osimertinib on the development of the fetus are unknown, and there is potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with osimertinib, breastfeeding should be discontinued if the mother is treated with these agents.
* Grade ≥ 2 blurred vision, conjunctivitis, corneal ulcer, dry eye, or keratitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Stinchcombe, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Osimertinib
Started | 17
Completed | 2
Not Completed | 15
Not completed — Disease Progression | 11
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Decline in Performance Status (PS) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Osimertinib
Number analyzed (Participants) | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [62 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
ECOG performance status [Count of Participants; unit: Participants] — All participants had an ECOG (Eastern Cooperative Oncology Group) score of 0 or 1. 0 = Fully active, able to carry on all pre-disease performance without restriction and 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    ECOG = 0 | 7
    ECOG = 1 | 10
EGFR mutation subtype [Count of Participants; unit: Participants] — EGFR = Epidermal growth factor receptor
  Participants
    G719X | 7
    L861Q | 6
    G719X/L718X | 1
    G719X/S768I | 1
    L861Q/S768I | 1
    G719X/V689L | 1
Location of metastases [Count of Participants; unit: Participants] — Participants could have more than one location for metastases.
  Participants
    Bone | 8
    Brain | 5
    Liver | 5
    Lung | 4
    Lymph node | 8
    Pleura | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate as Assessed by the Investigator Using Response Evaluation Criteria In Solid Tumors (RECIST 1.1)
Description: The number of participants who have a partial response or complete response to the study drug. Complete response (CR) = Disappearance of all target lesions and reduction in the short axis measurement of all pathologic lymph nodes to ≤10 mm; partial response (PR) = ≥30% decrease in the sum of the longest diameter of the target lesions compared with baseline.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 17
Participants | 8

2. Secondary Outcome: Progression Free Survival (PFS) as Measured by Response Evaluation Criteria In Solid Tumors (RECIST 1.1)
Description: Progression will be defined as time from starting study therapy to disease progression or death (whichever occurs first).
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Osimertinib
Number analyzed (Participants) | 17
months | 10.5 [5.0 to 15.2]

3. Secondary Outcome: Number of Participants With Adverse Events (AEs) as Measured by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Description: Adverse events (regardless of attribution) observed in all enrolled participants, except for those withdrawn prior to study treatment or fail to receive study treatment for various reasons. Counts and percentages of participants who experienced any AEs are calculated.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 17
Participants
  Diarrhea | 13
  Fatigue | 9
  Anorexia | 7
  Weight loss | 7
  Dyspnea | 6
  Vomiting | 5
  Abdominal pain | 5
  Cough | 4
  Acneiform rash | 4
  Maculopapular Rash | 4
  Respiratory failure | 1
  Thromboembolic event | 1

4. Secondary Outcome: Overall Survival as Noted by Follow-up Via Composite of Telephone or Medical Record Review.
Description: Overall survival as defined as time from starting study therapy until death from any causes.
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Osimertinib
Number analyzed (Participants) | 17
months | 13.8 [9.3 to 29.2]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Osimertinib
All-Cause Mortality (participants affected / at risk) | 12/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib (N=17)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib (N=17)
Diarrhea (Gastrointestinal disorders) | 13
Fatigue (General disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 7
Weight loss (Metabolism and nutrition disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Abdominal pain (General disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Acneiform rash (Skin and subcutaneous tissue disorders) | 4
Maculopapular rash (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03434418/Prot_SAP_000.pdf